CLINICAL TRIAL: NCT04939454
Title: Involvement of Skeletal Muscle Fibrocytes in sarcOpenia in Patients With Chronic ObstRuctive Pulmonary Disease
Acronym: MOTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2020/50
Record Dates: First submitted 2021-06-11; First posted 2021-06-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is an observational, etiological, cross-sectional case-control type, monocentric, multi-departmental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sarcopenic COPD patient (Experimental)
  Interventions: Procedure: quadricipital biopsy
- non-sarcopenic COPD patient (Other)
  Interventions: Procedure: quadricipital biopsy

INTERVENTIONS:
Procedure: quadricipital biopsy — The primary endpoint will be evaluated by histological examination only. The technique of percutaneous biopsy using the modified Bergström needle technique is currently considered the best alternative in the context of research, as it allows sufficient material to be obtained for various analyses and is much less invasive than the reference technique (surgical biopsy). Indeed, unlike surgical biopsy which requires an operating room and is a relatively heavy procedure (two suture planes, skin incision of several centimeters, resting for 48 hours after the procedure...), percutaneous biopsy by the modified Bergström technique can be performed in a consultation room, requires only one stitch, and allows resumption of walking 30 minutes after the end of the procedure.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is presently the third leading cause of death worldwide and is characterized by irreversible airflow limitation diagnosed by spirometry. COPD is currently considered as a systemic disease with predominantly respiratory involvement, associated with numerous comorbidities. Among these, muscle wasting, present in about one third of patients, is associated with a higher mortality (up to 10-fold, irrespective of the severity of the obstruction). Muscle wasting is classically characterized by a decrease in muscle strength and volume (sarcopenia), which can be defined by a decrease in the muscle mass measured by dual X-ray absorptiometry: Appendicular Skeletal Muscle Mass or ASM / height < 7.0 kg/m2 in men and 5.5 kg/m2 in women. However, sarcopenia is largely underestimated in current clinical practice. Moreover, there is no specific treatment: only exercise training as part of respiratory rehabilitation has shown some efficiency. The underlying pathophysiological mechanisms are indeed poorly characterized.

Fibrocytes, cells derived from blood monocytes and able to migrate to different organs in order to play pro-fibrotic or pro-inflammatory roles, play a key role in bronchial obstruction. They are recruited in the blood of COPD patients during an acute exacerbation according to a CXCL12/CXCR4 chemotactic axis. Their role in COPD sarcopenia is currently unknown, but recent data show that they are involved in a mouse model of muscular dystrophy.

The hypothesis is that fibrocytes are involved in COPD sarcopenia.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common and potentially serious chronic inflammatory respiratory disease. It has an estimated prevalence of 12% in Europe, making it a major public health issue. It is currently the third leading cause of death worldwide and affects a higher proportion of men (sex ratio 1.5:1.9). The main risk factor is cigarette smoke exposure (whether active or passive), responsible for 80% of cases. Exposure to other agents such as fine particles and fuel smoke can also lead to the development of the disease. Finally, a favourable genetic background is now commonly accepted as a risk factor.

COPD diagnosis is based on lung function measurement : non-reversible obstructive respiratory syndrome, i.e. a Tiffeneau coefficient (FEV1/FVC) < 70% after inhalation of a bronchodilator agent. At the pulmonary level, it is characterized by bronchial remodeling associated with parenchymal destruction, resulting on the one hand in peribronchial fibrosis, and on the other hand in emphysema bullae related to the rupture of the alveolar walls.

Its management is global and combines a series of medicinal and non-medicinal measures: use of bronchodilators and inhaled corticosteroids, smoking cessation (if applicable), prevention strategies including vaccination, physical management such as respiratory rehabilitation and management of comorbidities.

Indeed, COPD is currently considered a systemic disease with predominantly respiratory involvement associated with numerous comorbidities. These include cardiovascular disease, osteoporosis, depression, bronchopulmonary cancer and muscle dysfunction. The latter is characterized by a decrease in muscle strength and volume and is also called sarcopenia. Sarcopenia is present in 4 to 66% of patients and is associated with a particularly severe patient profile, since patients with low muscle mass have a mortality 13 times higher than patients with normal muscle mass (after adjustment for respiratory function).

Sarcopenia is defined by the loss of both muscle mass and strength, and extensive work has been done in the geriatric population, leading to the drafting of European recommendations which are considered applicable in the COPD population. Thus, sarcopenia can be defined by a decrease in the appendicular muscle mass index (ASM or Appendicular Skeletal Muscle Mass divided by height) measured by dexametry (or biphotonic X-ray absorptiometry), of less than 7.0 kg/m2 in men and 5.5 kg/m2 in women. However, although the measurement of lean body mass is recommended by both the HAS (COPD care pathway guide) and the latest recommendations of the Société de Pneumologie de Langue Française (French language lung society), this condition is currently largely under-diagnosed in COPD patients. Moreover, there is no specific treatment for sarcopenia: the only intervention that has been shown to be effective is exercise training as part of respiratory rehabilitation.

Numerous studies have described the histological changes characterizing muscle damage in COPD patients, particularly in the quadriceps. These include a decrease in the diameter and vascularization of muscle fibers, associated with a change in fiber metabolism: disappearance of type I fibers (predominantly oxidative metabolism) in favor of type II fibers (glycolytic metabolism). Local inflammation is also observed, sometimes associated with necrosis and an increase in the percentage of regenerating fibers. However, the originating mechanisms are still largely unknown.

Fibrocytes are cells derived from blood monocytes and able to migrate from the blood flow to different organs. They can exert pro-fibrotic functions by secreting collagen themselves or activating collagen secretion by fibroblasts. This is notably the case in the lung of COPD patients, where they play a key role in bronchial obstructive disease: they are recruited in the blood during an acute exacerbation of COPD, and their density is increased at the peribronchial level and negatively correlated with the parameters of lung function.

However, they may also play a pro-inflammatory role and influence the metabolism of resident cells. It has recently been shown that their differentiation is accompanied by a metabolic reprogramming that promotes oxidative phosphorylation. Moreover, recent data obtained in a mouse model show their involvement in tissue repair after muscle injury.

Because of their capacity to secrete pro-inflammatory factors and their possible influence on the metabolism of myofibers, studying their role in the development of sarcopenia in COPD patients could therefore be a promising avenue. Moreover, due to their preferential recruitment via a CXCL12/CXCR4 chemotactic axis, the migration of these cells towards damaged tissues (lung, muscle) of COPD patients would potentially respond to a therapeutic strategy by CXCR4 modulation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 40 years of age or older;
* Diagnosed with COPD according to the 2018 Global Initiative for Lung Disease (GOLD) criteria:

  * Smoking intoxication greater than or equal to 10 pack-years
  * Bronchial obstruction on spirometry with a FEV1 to FVC ratio post-bronchodilator < 70%.
* Available measurement of lean body mass by bioelectrical impedancemetry performed as part of routine care;
* Insured under the French social security system;
* Informed consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

The patients included will be sarcopenic and non-sarcopenic (equal numbers in each group, patients categorized according to the result of dexametry), and will be matched on sex and age (± 5 years).

Exclusion Criteria:

* Other concomitant respiratory pathology (e.g., asthma);
* Acute exacerbation of COPD or acute intercurrent condition (e.g. infection) ongoing or resolved within the last 48 hours
* Current systemic corticosteroid therapy;
* Contraindication to muscle biopsy: acquired or innate hemostasis disorders, anticoagulant therapy or double anti-platelet aggregation; contraindication to lidocaine: known hypersensitivity, patients with recurrent porphyrias;
* Presence of a concomitant muscular pathology, innate (e.g. genetic myopathy) or acquired (e.g. myositis);
* Progressive bronchopulmonary cancer;
* Pregnant or breast-feeding woman;
* Patient undergoing respiratory rehabilitation;
* Refusal to participate in the study.

Exclusion criteria between V1 and V2:

* Disorders of hemostasis detected on the blood sample;
* Pregnancy in progress.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Fibrocytes density (number/mm2) in quadricipital biopsies of sarcopenic patients versus non-sarcopenic patients | Day 14
  Fibrocytes density (number/mm2) in quadricipital biopsies of sarcopenic patients versus non-sarcopenic patients

SECONDARY OUTCOMES:
Mesure of appendicular skeletal muscle mass index (kg/m2) | Day 7
  Correlation between quadricipital fibrocytes density and appendicular skeletal muscle mass index (kg/m2)
Distance covered in 6 minutes (meters) | Day 7
  Correlation between quadricipital fibrocytes density and parameters evaluating muscular function (handgrip test, mid-thigh cross-sectional area, impedance ratio and phase angle in bioelectrical impedance, quadriceps sonographic echogenicity...)
Maximum grip forces with hand dynamometer in kg | Day 7
  Correlation between quadricipital fibrocytes density and parameters evaluating muscular function (handgrip test, mid-thigh cross-sectional area, impedance ratio and phase angle in bioelectrical impedance, quadriceps sonographic echogenicity...)
Average of the maximum forces developed in isokinetic dynamometry for the quadriceps in N.m-1 | Day 7
  Correlation between quadricipital fibrocytes density and parameters evaluating muscular function (handgrip test, mid-thigh cross-sectional area, impedance ratio and phase angle in bioelectrical impedance, quadriceps sonographic echogenicity...)

CONTACTS AND LOCATIONS:
Overall Officials: Pauline HENROT, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Hôpital Haut-Lévêque - CHU de Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No